CLINICAL TRIAL: NCT06793982
Title: The Efficacy of Platelet Rich Plasma Compared With Corticosteroid Injections for the Treatment of Pain Associated With Hip Osteoarthritis
Brief Title: Platelet Rich Plasma Versus Corticosteroids in Hip Osteoarthritis Pain
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: LifeBridge Health (Other)
Collaborators: Hip Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2084137
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Hip Osteoarthritis
Keywords: platelet rich plasma; hip osteoarthritis; PRP; hip OA; Corticosteroids
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant
Masking Description: Given the nature of this study, blinding will not be possible for the treating surgeon and research staff. The participants will be blinded from the regimen that they receive, and both groups will have blood drawn and the injection will be covered in a manner to ensure participants cannot ascertain the treatment regimen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Autologous Platelet Rich Plasma (Experimental): ~Injection of approximately 10 mL autologous PRP Magellan Autologous Concentration System, ISTO Biologics
  Interventions: Device: Platelet Rich Plasma Joint Injection
- Corticosteroid (Active Comparator): 5 milliliters (mL) injection of corticosteroid (1cc Kenalog, 4cc Xylocaine) Kenalog - 40 (triamcinolone acetonide injectable suspension, USP) Xylocaine - MPF (lidocaine HCl Injection, USP)
  Interventions: Drug: Corticosteroid Injection

INTERVENTIONS:
Device: Platelet Rich Plasma Joint Injection — Magellan Autologous Concentration System, ISTO Biologics
  Arms: Autologous Platelet Rich Plasma
Drug: Corticosteroid Injection — 5 milliliters (mL) injection of corticosteroid (1cc Kenalog, 4cc Xylocaine) Kenalog - 40 (triamcinolone acetonide injectable suspension, USP) Xylocaine - MPF (lidocaine HCl Injection, USP)
  Arms: Corticosteroid

SUMMARY:
Prospective, single-center that may go on to being multicenter, randomized trial comparing platelet rich plasma (PRP) versus corticosteroid injection for the treatment of symptoms of Hip osteoarthritis. The purpose of the study is to determine which therapy provides a greater reduction in patient reported outcome measures of pain and function.

DETAILED DESCRIPTION:
Platelet rich plasma has become increasingly utilized as a treatment option for Hip osteoarthritis. Corticosteroids is currently an approved medication to treat the symptoms of the Hip osteoarthritis. There is limited evidence in a prospective randomized manner powered adequately to determine a difference between these treatments for pain associated with Hip osteoarthritis.

Prospective, single center that may go on to be multi-center, single blind (participant), randomized trial comparing platelet rich plasma (PRP) versus corticosteroid injection for the treatment of symptoms of Hip osteoarthritis. The purpose of the study is to determine which therapy provides a greater reduction in patient reported outcome measures of pain and function.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 21-80 years
* Radiographic diagnosis of Kellgren-Lawrence (KL) grade of II or III Hip osteoarthritis
* Indicated for a Hip injection to treat Hip OA symptoms

Exclusion Criteria:

* Any injections into the target Hip within three months
* Current overlying skin infection
* Current or previous diagnosis of "chronic pain"
* Opioid tolerant at time of screening (for a week or longer, at least 60 mg of morphine daily, or at least 30 mg of oral oxycodone daily, or at least 8 mg of oral hydromorphone daily or an equianalgesic dose of another opioid.)
* Allergy to any potential ingredients or medications utilized in any of the two groups
* Treatment with another investigational drug or other intervention for pain
* Diagnosis of Diabetes Mellitus
* If female, pregnant or planning to be pregnant within the following 3 months or study duration
* Any condition(s) or diagnosis, both physical or psychological, or physical exam finding in the opinion of the investigator that would precludes participation

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain Score VAS | baseline, six weeks, and three months
  Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10 cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). Pain intensity that is calculated by measuring the distance from the "no pain" end of a line to a mark placed by the patient to indicate their current pain level. This will be measured at baseline, six weeks, and three months.

SECONDARY OUTCOMES:
Pain Score NRS | baseline, six weeks, and three months.
  Numeric Pain Rating Scale (NRPS) where patients are asked to rate their pain on a scale of 0 to 10, with 0 representing "no pain" and 10 representing "the worst pain imaginable. This will be measured at baseline, six weeks, and three months.
Functional score HOOS | baseline, six weeks, and three months
  The hip disability and osteoarthritis outcome score (HOOS) is a questionnaire intended to be used to assess patient's opinions about their hip and associated problems and to evaluate their symptoms and functional limitations during a therapeutic process. The HOOS includes 40 items with five possible responses, graded from 0 to 4 (0 points = worst possible score; 100 points = best possible score). Standardized answer options are given in 5 Likert boxes with scores from 0 to 4 (no, mild, moderate, severe and extreme) to answer the questions. This will be measured at baseline, six weeks, and three months.
Functional score HHS | baseline, six weeks, and three months
  The Harris Hip Scale (HHS) was developed for the assessment of the results of hip surgery, and is intended to evaluate various hip disabilities and methods of treatment in an adult population. The maximum score possible is 100. Results can be interpreted with the following[1]: <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent. This will be measured at baseline, six weeks, and three months.
Functional score WOMAC | baseline, six weeks, and three months
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright. The total WOMAC score is the sum of the three subscale scores, with a possible score range of 0-96. Higher scores indicate worse pain, stiffness, and functional limitations. This will be measured at baseline, six weeks, and three months.
Pain Medication Adherence | Baseline through three months
  Measured by number of days until pain medication (acetaminophen) is not adequate.

CONTACTS AND LOCATIONS:
Locations (1):
- Sinai Hospital of Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No